CLINICAL TRIAL: NCT05736523
Title: Improving Early Detection of Melanoma Recurrence With Circulating Tumor DNA (ctDNA)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Intermountain Medical Center (Other); Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 133519
Record Dates: First submitted 2022-09-16; First posted 2023-02-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: Stage II Melanoma; Stage III Melanoma; ctDNA; Circulating Tumor DNA; surgical resection; tumor marker; melanoma recurrence
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both tumor, from FFPE blocks, and blood will be collected, processed and tested. Whole blood samples will be taken within 4 weeks prior to complete surgical resection of the primary tumor and sentinel nodes. Separate samples will be drawn postoperatively within 4 weeks after full resection of all known disease and every 3-6 months following for 3 years post-surgery. All blood samples will be sent for ctDNA testing. Primary tumor tissue (FFPE) will be collected and sent with initial blood sample to lab for ctDNA testing. If available, additional primary tumor tissue will be banked for future nucleic acid extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-randomized experimental biomarker study evaluating ctDNA levels in patients with stage IIB/C and stage IIIB/C/D melanoma skin cancer pre and post-surgery

Study participants will complete a ctDNA test within 4 weeks of their planned surgical resection of their melanoma. Within 4 weeks post-surgery another ctDNA test will be completed. During these time points stool samples and diet questionnaires will be collected for biospecimen banking.

DETAILED DESCRIPTION:
The investigators hypothesize that ctDNA levels drawn before and after surgical resection of a primary tumor and either sentinel lymph nodes or clinically involved metastatic lymph nodes will correlate with the presence of sentinel node microscopic metastatic disease and clinically evident nodal metastatic disease. The investigators also predict that approximately 20% of sentinel lymph node negative Stage IIB/IIC patients will have evidence of ctDNA positivity post-surgery.

Primary Objective:

* To assess the feasibility of generating patient specific ctDNA assay from Signatera© test for primary melanoma samples submitted with clinical stage IIB/IIC and stage III melanoma patients.

Secondary Objective(s):

* To investigate serum levels of melanoma ctDNA pre and postoperatively in clinical Stage IIB/C and Stage III melanoma patients.
* To evaluate the relationship of serum ctDNA levels pre-operatively with sentinel lymph node biopsy status in clinical Stage IIB/C patients.
* Evaluate for clearance or persistence of ctDNA levels post complete resection in patients with clinically evident lymph node metastasis (Stage IIIB/C/D).
* Assess feasibility of collection of pre- and post-operative stool samples

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient must be ≥ 18 years of age.
* Patient must be a surgical candidate with Stage IIB, IIC melanoma or fully resectable Stage III B/C/D cutaneous melanoma.
* Patients with resectable in transit/nodal metastatic disease who have had prior adjuvant or systemic/intralesional therapy can be included provided that the planned resected lesions either progressed or developed while on or after completion of prior treatment. Patients with resectable in transit/nodal metastatic disease who are treated with neoadjuvant therapy prior to resection are also eligible provided that the initial blood and tumor biopsy sample are taken prior to initiation of neoadjuvant therapy.
* Tissue available meeting one of the following criteria:

  1. For patients with Clinical stage II primary tumors that have been biopsied prior to evaluation by the surgeon, or those with stage III tumors that have been partially/fully excised prior to definitive surgery, adequate tissue will be confirmed prior to enrollment to follow Natera's tissue sample collection instructions when selecting the appropriate specimen.

     OR
  2. For patients with bulky lymph nodes involved with clinically evident, biopsy proven metastatic disease, in transit metastasis, or with extensive residual primary tumor present prior to excision, and in the treating surgeon's assessment there will be extensive tumor for evaluation, the patient can be enrolled with tissue adequacy evaluation post resection
* Patient is willing to provide blood samples for Signatera testing as outlined in the study calendar.
* Patient is able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

EXCLUSION CRITERIA:

* Patient is unable to provide informed consent or is unwilling to sign an approved consent form.
* Patient has other clinically significant disorders that would preclude safe study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who have Stage IIB/C or Stage IIB/C/D melanoma skin cancer
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Serum ctDNA acquisition, processing and results | Within 4 weeks pre-surgery through a maximum of 4 weeks post-surgery
  The proportion of cases in which sample acquisition, processing and return of results from the two initial ctDNA (serum VAF allele levels, ng/ml) analyses occurs within 6 weeks of acquisition of the post-operative serum sample. The two ctDNA analyses are from the initial tumor biopsy and blood, and post-operative blood draw.

SECONDARY OUTCOMES:
Pre and Post-operative Serum Variant Allele Frequency | Within 4 weeks pre-surgery through a maximum of 4 weeks post-surgery
  Pre-operative and post-operative serum Variant allele frequency (VAF) ng/ml from the Signatera© test in all evaluable patients
Association of pre-operative and post-operative serum Variant allele frequency (VAF) levels (ng/ml) from the Signatera© test and sentinel lymph node biopsy metastatic status | Within 4 weeks pre-surgery
  Evaluate the relationship of serum Variant allele frequency (VAF) levels (ng/ml) pre-operatively with sentinel lymph node biopsy clinical outcome (positive/negative for metastatic disease) in clinical Stage IIB/C melanoma patients undergoing sentinel lymph node biopsy.
Pre-operative serum VAF levels (ng/mL) from Signatera© stratified by pre-operative sentinel lymph node and clinically evident lymph node metastatic status. | Within 4 weeks post-surgery
  Evaluate association of pre-operative serum VAF levels (ng/ml) from Signatera© stratified by pre-operative sentinel lymph node eligible (Clinical stage IIB/IIC) patients vs. patients with clinically evident lymph node metastases (clinical stage III).
Quantify the number of patients who develop detectable VAF levels (ng/ml) within the first 3 years after surgery and evaluate possible correlation with recurrence. | 3 years post resection of the last patient enrolled.
  Proportion of participants with detectable VAF levels (ng/ml) using the Signatera© test at any time point during the surveillance period and any clinical or radiologic evidence of recurrence.
Pre and Post-operative Stool Samples | Within 4 weeks pre-surgery through a maximum of 4 weeks post-surgery
  Proportion of cases in which pre-operative and post-operative patient stool samples are successfully obtained
The proportion of patients for which serum VAF levels (ng/ml) are undetectable post complete resection of either sentinel nodes or clinically evident lymph node metastases | Within 4 weeks post-surgery
  The proportion of patients for which serum VAF levels (ng/ml) are undetectable post complete resection of either sentinel nodes or clinically evident lymph node metastases

CONTACTS AND LOCATIONS:
Overall Officials: John Hyngstrom, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Background] Gershenwald JE, Scolyer RA, Hess KR, Sondak VK, Long GV, Ross MI, Lazar AJ, Faries MB, Kirkwood JM, McArthur GA, Haydu LE, Eggermont AMM, Flaherty KT, Balch CM, Thompson JF; for members of the American Joint Committee on Cancer Melanoma Expert Panel and the International Melanoma Database and Discovery Platform. Melanoma staging: Evidence-based changes in the American Joint Committee on Cancer eighth edition cancer staging manual. CA Cancer J Clin. 2017 Nov;67(6):472-492. doi: 10.3322/caac.21409. Epub 2017 Oct 13. PMID 29028110
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Long GV, Hauschild A, Santinami M, Atkinson V, Mandala M, Chiarion-Sileni V, Larkin J, Nyakas M, Dutriaux C, Haydon A, Robert C, Mortier L, Schachter J, Schadendorf D, Lesimple T, Plummer R, Ji R, Zhang P, Mookerjee B, Legos J, Kefford R, Dummer R, Kirkwood JM. Adjuvant Dabrafenib plus Trametinib in Stage III BRAF-Mutated Melanoma. N Engl J Med. 2017 Nov 9;377(19):1813-1823. doi: 10.1056/NEJMoa1708539. Epub 2017 Sep 10. PMID 28891408
- [Background] Weber J, Mandala M, Del Vecchio M, Gogas HJ, Arance AM, Cowey CL, Dalle S, Schenker M, Chiarion-Sileni V, Marquez-Rodas I, Grob JJ, Butler MO, Middleton MR, Maio M, Atkinson V, Queirolo P, Gonzalez R, Kudchadkar RR, Smylie M, Meyer N, Mortier L, Atkins MB, Long GV, Bhatia S, Lebbe C, Rutkowski P, Yokota K, Yamazaki N, Kim TM, de Pril V, Sabater J, Qureshi A, Larkin J, Ascierto PA; CheckMate 238 Collaborators. Adjuvant Nivolumab versus Ipilimumab in Resected Stage III or IV Melanoma. N Engl J Med. 2017 Nov 9;377(19):1824-1835. doi: 10.1056/NEJMoa1709030. Epub 2017 Sep 10. PMID 28891423
- [Background] Christensen E, Birkenkamp-Demtroder K, Sethi H, Shchegrova S, Salari R, Nordentoft I, Wu HT, Knudsen M, Lamy P, Lindskrog SV, Taber A, Balcioglu M, Vang S, Assaf Z, Sharma S, Tin AS, Srinivasan R, Hafez D, Reinert T, Navarro S, Olson A, Ram R, Dashner S, Rabinowitz M, Billings P, Sigurjonsson S, Andersen CL, Swenerton R, Aleshin A, Zimmermann B, Agerbaek M, Lin CJ, Jensen JB, Dyrskjot L. Early Detection of Metastatic Relapse and Monitoring of Therapeutic Efficacy by Ultra-Deep Sequencing of Plasma Cell-Free DNA in Patients With Urothelial Bladder Carcinoma. J Clin Oncol. 2019 Jun 20;37(18):1547-1557. doi: 10.1200/JCO.18.02052. Epub 2019 May 6. PMID 31059311
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Background] Iafolla, Marco & Yang, SY Cindy & Dashner, Scott & Xu, Wei & Hansen, Aaron & Bedard, Philippe & Lheureux, Stéphanie & Spreafico, Anna & Razak, Albiruni & Wu, Hsin-Ta & Shchegrova, Svetlana & Liu, Zhihui & Ohashi, Pamela & Torti, Dax & Louie, Maggie & Sethi, Himanshu & Aleshin, Alexey & Siu, Lillian & Bratman, Scott & Pugh, Trevor. (2019). Bespoke circulating tumor DNA (ctDNA) analysis as a predictive biomarker in solid tumor patients (pts) treated with single-agent pembrolizumab (P).. Journal of Clinical Oncology. 37. 2542-2542. 10.1200/JCO.2019.37.15_suppl.2542.
- [Background] Magbanua, MJM & Swigart, Lamorna & Hirst, Gillian & Yau, C & Wolf, Denise & Ma, AA & Bergin, E & Venters, S & Sethi, H & Wu, H-T & Tin, Tony & Sawyer, S & Louie, M & Zimmermann, Bernhard & Lin, C-HJ & Keats, J & Liang, WS & (Phillips) Cuyugan, Lori & van 't Veer, Laura. (2019). Abstract PD2-01: Personalized serial circulating tumor DNA (ctDNA) analysis in high-risk early stage breast cancer patients to monitor and predict response to neoadjuvant therapy and outcome in the I-SPY 2 TRIAL. Cancer Research. 79. PD2-01. 10.1158/1538-7445.SABCS18-PD2-01.
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Mounessa JS, Caravaglio JV, Dellavalle RP. Comparison of Regional and State Differences in Melanoma Rates in the United States: 2003 vs 2013. JAMA Dermatol. 2017 Mar 1;153(3):345-347. doi: 10.1001/jamadermatol.2016.4625. No abstract available. PMID 28030665
- See also: Signatera Advanced Cancer Detection | Natera — https://www.natera.com/signatera
- See also: U.S. Cancer Statistics Working Group. U.S. Cancer Statistics Data Visualizations Tool, — https://www.cdc.gov/cancer/dataviz